CLINICAL TRIAL: NCT03362970
Title: Improvements Through the Use of a Rapid Multiplex PCR Enteric Pathogen Detection Kit in Children With Hematochezia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: REB17-1916
Record Dates: First submitted 2017-11-21; First posted 2017-12-05 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2022-05

CONDITIONS: Diarrhea Bloody
Keywords: Bloody Diarrhea; STEC; Hematochezia; BioFire FilmArray; Child
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data extractors and Investigators will be unaware of allocation assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (Active Comparator): For children randomized to the standard of care arm, the treating physician will be informed to proceed as per their usual practice and treatment patterns. If stool is unavailable a rectal swab will be collected and sent to Calgary Laboratory Services (CLS) for routine culture. A routine stool specimen for back-up culture will still be requested as per standard of care. Home stool collection will be performed for those unable to provide a sample at enrolment and will be achieved by providing families with collection kits.
  Interventions: Other: Standard of Care
- BioFire Gastrointestinal Panel FilmArray (Experimental): For children randomized to the BioFire FilmArray arm, stool, if available, will be sent STAT to Calgary Laboratory Services (CLS) for the performance of the BioFire FilmArray test and routine culture. If stool is unavailable, a rectal swab will be performed and sent to CLS for the performance of the BioFire FilmArray test and routine culture. A routine stool specimen for back-up culture will still be requested as per standard of care once it is available. Treatment decisions will be at the sole discretion of the ED treating physician who receives the result.
  Interventions: Device: BioFire Gastrointestinal Panel FilmArray®

INTERVENTIONS:
Device: BioFire Gastrointestinal Panel FilmArray® — The BioFire Gastrointestinal Panel FilmArray® is a multiplexed nucleic acid (NA) based device that simultaneously identifies 22 enteric pathogens. It specifically tests for the presence of Shiga toxin and for O157. It requires 2 minutes of hands-on-time, returns results in ~2-3 hour, and is Health Canada and Food and Drug Administration approved. The device, which has been validated, hopefully will enable the early identification of infected children and initiation (or withholding) of interventions directed by previously unavailable clinical data. It will enable us to bring a precision medicine approach into ED care.
  Arms: BioFire Gastrointestinal Panel FilmArray
Other: Standard of Care — Standard practices for children with hematochezia upon the discretion of the treating physician. If investigations are ordered, results have a turn-around time up to 72 hours.
  Arms: Standard of Care

SUMMARY:
Children presenting for emergency department (ED) care with bloody diarrhea (i.e. hematochezia) represent a diagnostic challenge. Infectious enteric pathogens - Salmonella, Shigella and Shiga toxin-producing Escherichia coli (STEC) - are at the top of the differential diagnosis list. STEC is of greatest concern because ~15% of infected children develop the Hemolytic Uremic Syndrome (HUS). Our team has demonstrated that antibiotic administration to STEC-infected children increases the risk of developing HUS while dehydration is associated with mortality. Rapidly identifying children with STEC infection can reduce unnecessary resource use in uninfected children while providing them to those with confirmed STEC infection. The study team will conduct a prospective ED-based study that will randomly allocate 60 children to either standard care as dictated by the treating physician or to the use of a 22-pathogen, nucleic acid based, 1-hour run time diagnostic test. The study team will evaluate the impact of testing on clinical resource use, clinical outcomes, costs and patient satisfaction.

DETAILED DESCRIPTION:
Background:

The rapid identification of STEC-infected children will enable the provision of appropriate and timely care to such children. The rapid identification of other enteric pathogens (bacteria, virus, parasite) will enable the provision of targeted therapies as appropriate and the withholding of avoidable interventions. It will also provide information for clinicians to consider alternate, non-infectious etiologies as appropriate. The study team hypothesize that the BioFire FilmArray can be used selectively in children with hematochezia to identify children with STEC infection and therefore will expeditiously identify children in need of therapeutic interventions and those for whom blood testing, intravenous fluids, and follow-up visits are unnecessary. Knowledge of the etiology early in the course of disease will enhance the provision of a patient-level precision medicine approach to what is otherwise an ill-defined symptom.

Study Design:

The study team will prospectively identify children who present with hematochezia. Potentially eligible subjects will be identified by our Pediatric Emergency Medicine Research Associate Program (PEMRAP) and the Pediatric Emergency Research Team (PERT) nurses (ED coverage 14 hours per day). Eligible children will have ≥3 episodes of diarrhea within the preceding 24 hours and will have had blood identified in the stool (by physician, nurse or parent ). Eligible subjects will be approached by a PERT team member to obtain consent (and assent when appropriate). Once consent has been obtained, study participants will be randomized by a REDCap randomization tool to ensure allocation concealment (i.e. research team, ED physicians will be unaware until after enrolled into the study and randomized).

Children randomized to the standard of care arm will have demographic and clinical information collected and the treating physician will be informed to proceed as per their usual practice and treatment patterns. If stool is unavailable a rectal swab will be collected and sent to Calgary Laboratory Services (CLS) for routine culture. A routine stool specimen for back-up culture will still be requested as per standard of care. Home stool collection will be performed for those unable to provide a sample at enrolment and will be achieved by providing families with collection kits. Sample specimens may be stored at CLS as per routine procedures for standard clinical care. Following the completion of the visit, data regarding all testing, procedures, and medications administered will be collected. The family will be contacted 14 days later to collect outcome information (clinical and health resource use) and satisfaction. The medical records and select administrative databases may be reviewed to ascertain and confirm outcome data on Day 28.

Children randomized to the BioFire FilmArray arm will have the same data collected, but stool, if available, will be sent STAT to Calgary Laboratory Services (CLS) for the performance of the BioFire FilmArray test and routine culture. If stool is unavailable, a rectal swab will be performed and sent to CLS for the performance of the BioFire FilmArray test and routine culture. A routine stool specimen for back-up culture will still be requested as per standard of care once it is available. Sample specimens may be stored at CLS as per routine procedures for standard clinical care. The result of the BioFire test will be printed and brought to the ED where it will be provided to the ED physician for immediate review and management as appropriate. The result will be included in the ED chart for documentation purposes. Education regarding the interpretation of BioFire FilmArray results will have been performed in advance to all faculty members and a research team member will be available to answer any questions should they arise. We have worked with leaders at CLS including Drs. Gregson, Berenger and Vanderkooi who believe we should be able to receive a result within 2-3 hours of receipt of the specimen at CLS. Treatment decisions will be at the sole discretion of the ED treating physician who receives the result. Following the completion of the visit, data regarding all testing, procedures, and medications administered will be collected. The family will be contacted 14 days later to collect outcome information (clinical and health resource use) and satisfaction. The medical records and select administrative databases may be reviewed to ascertain and confirm outcome data on Day 28.

For those who decline consent, the study team will request consent to access select administrative data, Netcare and/or access to the child's medical records related to the illness to document interventions and outcomes in order to be able to assess bias by comparing participating and non-participating children in this study.

Objectives:

Primary Objective

1. To determine if use of the BioFire FilmArray in children with hematochezia results in a reduction in resource utilization. Primary outcome - any blood tests (dichotomous with sub-analysis by specific blood tests); secondary - intravenous fluid administration, ED encounters.

Secondary Objectives

1. To quantify clinical outcomes - development of HUS, acute kidney injury, need for renal replacement therapy, turnaround time from BioFire result relative to stool culture result.
2. To determine if use of the BioFire FilmArray is associated with greater family satisfaction with care.
3. To determine testing criteria to optimize the clinical improvement emerging from use of the BioFire FilmArray (i.e. predictors of bacterial etiology).

Significance:

The study team intend to determine new knowledge:

1. If use of the BioFire FilmArray, a rapid, multi-analyte enteric pathogen detection device, reduces resource utilization in a pediatric ED when employed on children with bloody diarrhea. The study team hypothesize that use of the test combined with behavioural changes by physicians will reduce the use of baseline blood tests, the administration of intravenous fluids and future health-care resource use (children are often brought back for repeat blood tests and fluids while awaiting culture results).
2. If satisfaction is higher in individuals randomized to testing with the BioFire FilmArray arm compared with children in the standard care arm.

Potential child health improvements:

1. Children with STEC infection will be rapidly identified: The study team has shown that in the 2014 STEC outbreak in Alberta, the median time from initial health care presentation to stool sample collection was 7 hours (IQR 2, 28) and to sample receipt at the laboratory was 33 hours (IQR 18, 42). Even more concerning is that the time from initial health care encounter to positive culture was 120 (IQR 86, 205) hours. By collecting rectal swabs at the point of care, the study team will initiate specimen processing an average of 30 hours earlier. By employing the BioFire FilmArray the study team will reduce stool processing time by over 80 hours.
2. Children with STEC infection will have dehydration reversed rapidly and they will be closely monitored: Following the rapid identification of children with STEC infection, all such children will be managed in accordance with a protocol developed by the APPETITE team for Alberta Health Services (http://www.albertahealthservices.ca/assets/info/hp/diseases/if-hp-dis-ecoli-stec.pdf), which includes the performance and monitoring of serum biochemistry and hematologic profiles and the prevention of dehydration. It is believed that the early administration of intravascular volume expansion has the potential to reduce the morbidity of HUS in affected children. [Ake et al., 2005 & Hickey et al., 2011]
3. Children who do not have STEC infection will avoid unnecessary blood tests, intravenous fluids and repeat visits: As ~10% of eligible children will have STEC infection, [Klein et al., 2006 & Klein et al., 2002] the routine performance of blood tests, administration of intravascular hydration, and frequent monitoring is unnecessary in the vast majority of children with hematochezia. As such, knowledge that a result will be rapidly available will enable clinicians to confidently discharge children without performing unnecessary procedures. Those who test positive can be recalled to the ED for the appropriate management.
4. Children will have alternative etiologies identified rapidly: The BioFire FilmArray will also enable the rapid identification of other pathogens, some of which will require immediate therapy such as Shigella sp., Clostridium difficile, and others that have public health implications such as Salmonella sp., and norovirus.
5. Children who do not have infectious gastroenteritis will be rapidly identified: Children with a negative BioFire FilmArray will also be identified. This would raise the suspicion for alternative etiologies.
6. Transmission will be reduced: The rapid identification of infected children has the potential to reduce spread, which is common and occurs early in the course of disease. Transmission might be reduced by separating infected index cases from their at risk siblings. [Werber et al., 2008]

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 6 months - 17.99 years of age
2. Have ≥3 episodes of diarrhea within the preceding 24 hours and have blood identified in the stool (by physician, nurse or parent)

Exclusion Criteria:

1. Previously enrolled in the study
2. Unavailable for Day 14 follow-up
3. Currently (most recent complete blood count) known to be neutropenic (Neutrophils <1000), or at high-risk of being neutropenic (receiving chemotherapy) at present
4. Blood work performed prior to enrollment
5. Known to be STEC positive (stool culture, PCT, or toxin)
6. Pre-existing diagnosis of IBD (Crohn's disease, Ulcerative Colitis)
7. Language barrier that prevents the ability to obtain informed consent and assent (when appropriate)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MDCM, MSc, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ake JA, Jelacic S, Ciol MA, Watkins SL, Murray KF, Christie DL, Klein EJ, Tarr PI. Relative nephroprotection during Escherichia coli O157:H7 infections: association with intravenous volume expansion. Pediatrics. 2005 Jun;115(6):e673-80. doi: 10.1542/peds.2004-2236. PMID 15930195
- [Background] Hickey CA, Beattie TJ, Cowieson J, Miyashita Y, Strife CF, Frem JC, Peterson JM, Butani L, Jones DP, Havens PL, Patel HP, Wong CS, Andreoli SP, Rothbaum RJ, Beck AM, Tarr PI. Early volume expansion during diarrhea and relative nephroprotection during subsequent hemolytic uremic syndrome. Arch Pediatr Adolesc Med. 2011 Oct;165(10):884-9. doi: 10.1001/archpediatrics.2011.152. Epub 2011 Jul 22. PMID 21784993
- [Background] Klein EJ, Boster DR, Stapp JR, Wells JG, Qin X, Clausen CR, Swerdlow DL, Braden CR, Tarr PI. Diarrhea etiology in a Children's Hospital Emergency Department: a prospective cohort study. Clin Infect Dis. 2006 Oct 1;43(7):807-13. doi: 10.1086/507335. Epub 2006 Aug 22. PMID 16941358
- [Background] Klein EJ, Stapp JR, Clausen CR, Boster DR, Wells JG, Qin X, Swerdlow DL, Tarr PI. Shiga toxin-producing Escherichia coli in children with diarrhea: a prospective point-of-care study. J Pediatr. 2002 Aug;141(2):172-7. doi: 10.1067/mpd.2002.125908. PMID 12183710
- [Background] Werber D, Mason BW, Evans MR, Salmon RL. Preventing household transmission of Shiga toxin-producing Escherichia coli O157 infection: promptly separating siblings might be the key. Clin Infect Dis. 2008 Apr 15;46(8):1189-96. doi: 10.1086/587670. PMID 18444854

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between June 15, 2018 through May 7, 2022 in the emergency department of the Alberta Children's Hospital located in Calgary, Alberta, Canada.
Period: Overall Study
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 31 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.9 [1.3 to 9.8] | 2.7 [1.5 to 5.2] | 3.7 [1.4 to 6.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 20 | 18 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Blood Test Performance
Description: Any blood testing performed within 72 hours of randomization.
Time Frame: Day 28 of the study after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
Participants | 18 | 17

2. Secondary Outcome: Intravenous Fluid Administration
Description: Children administered IV fluids identified by chart review.
Time Frame: Day 28 of the study after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
Participants | 12 | 11

3. Secondary Outcome: Total Physician Visits (ED and Non-ED)
Description: Children visiting additional health-care practitioners identified by chart review.
Time Frame: Day 28 of the study after baseline
Measure: Median (Inter-Quartile Range); unit: physician visits
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
physician visits | 1 [0 to 1] | 0 [0 to 1]

4. Secondary Outcome: ED Length of Stay
Description: ED length of stay during enrollment visit determined by chart review.
Time Frame: Day 28 of the study after baseline
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
hours | 4.2 [2.9 to 5.6] | 4.6 [3.6 to 5.7]

5. Secondary Outcome: Antibiotic Use
Description: Antibiotic use identified by chart review.
Time Frame: Day 28 of the study after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
Participants | 5 | 6

6. Secondary Outcome: Hospital and Intensive Care Unit Admission
Description: Hospitalization identified by chart review.
Time Frame: Day 28 of the study after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
Participants | 2 | 5

7. Secondary Outcome: Diagnostic Imaging Performed
Description: Diagnostic imaging performed identified by chart review.
Time Frame: Day 28 of the study after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
Participants | 2 | 4

8. Secondary Outcome: Hemolytic-Uremic Syndrome (HUS)
Description: Children with HUS identified by chart review.
Time Frame: Day 28 of the study after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

9. Secondary Outcome: Acute Kidney Injury
Description: Based on chart review in accordance with KDIGO guidelines.
Time Frame: Day 28 of the study after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

10. Secondary Outcome: Need for Renal Replacement Therapy
Description: Renal replacement therapy identified by chart review.
Time Frame: Day 28 of the study after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

11. Secondary Outcome: Caregiver and Patient Satisfaction
Description: Satisfaction of care received during ED visit answered in Day 14 follow-up form on a Likert scale. Caregivers were asked the following question: "Using any number from 0 to 10, where 0 is the worst care possible and 10 is the best care possible, what number would you use to rate your child's care during the emergency department visit (Day 0 - Enrollment visit)?" the scale does not have a name or specific construct beyond as detailed in the script that was used to ask the question. The range is from 0 (minimum) to 10 (maximum). There are no sub-scales. Higher values represent greater satisfaction.
Time Frame: Day 14 of the study after baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
Number analyzed (Participants) | 29 | 31
units on a scale | 9 [8 to 10] | 9 [8 to 10]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for while in the emergency department, which was a median of 4.6 hours (IQR: 3.4-5.6).
Description: Adverse event definition did not differ from cliniclatrials.gov definition
Arm/Group | Standard of Care | BioFire Gastrointestinal Panel FilmArray
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT03362970/Prot_SAP_000.pdf